CLINICAL TRIAL: NCT02816567
Title: Laparoscopic Surgery and Abdominal Compliance Factors Including Neuromuscular Blocking Agents
Brief Title: Laparoscopic Surgery and Abdominal Compliance
Acronym: COELIOCUR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA16045
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Patients Ongoing Elective Abdominal Laparoscopy
MeSH Terms: interventions — Propofol; Sufentanil; Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- NMBA group (Experimental)
  Interventions: Drug: propofol; Drug: NMBA - cisatracurium; Drug: sufentanil; Procedure: laparoscopic surgery
- placebo group (Placebo Comparator)
  Interventions: Drug: propofol; Drug: placebo - isotonic saline serum; Drug: sufentanil; Procedure: laparoscopic surgery

INTERVENTIONS:
Drug: propofol
Drug: NMBA - cisatracurium
  Arms: NMBA group
Drug: placebo - isotonic saline serum
  Arms: placebo group
Drug: sufentanil
Procedure: laparoscopic surgery

SUMMARY:
The objective of the study is to describe factors influencing abdominal compliance during laparoscopic surgery, including neuromuscular blocking agents (NMBA). The use of NMBA is randomized and blinded from the surgeons and the anesthesiologist. The abdominal compliance is measured by pressure/volume relationship.

DETAILED DESCRIPTION:
Background and rationale. Abdominal laparoscopic surgery is widely used. The meet good conditions, the surgeons need a large enough workspace. Carbonic gaz is insufflated in the intraperitoneal space but limited by the induced pressure which usually must not be above 15mm mercury (Hg) because of subsequent organ failures. The relationship between pressure and gaz volume insufflated defines the abdominal compliance (ΔV/ΔP).

The use of neuromuscular blocking agents (NMBA) is often used during abdominal laparoscopic surgery in order to reduce abdominal tonus, create a sufficient laparoscopic workspace hence improving abdominal compliance. However, considering good working conditions could be achieved by the use of NMBA, other factors could be considered like body weight, length, BMI, surgical abdominal history, parity.

Main objective : To compare the working surgical conditions and the pneumoperitoinea volume obtained during abdominal laparoscopic surgery with and without initial NMBA use.

Hypothesis: The use of NMBA improve the incidence of good surgical working conditions.

Study Design : Randomized blinded clinical trial. Two patients groups are compared, one receiving NMBA and one receiving a placebo. Randomisation will be realised by 1/1 ratio in blocks of 4.

The primary outcome is a composite criteria : the obtention of laparoscopic workspace greater than 3 liters associated with an abdominal pressure lesser than 15mmHg and a good surgical rating scale.

A statistical analysis reveal that 90 patients in each group need to be included from estimated 90% satisfying surgical conditions in NMBA group and 70% in placebo group.

In the placebo group, when surgical conditions are not correct (insufflated volume lesser than 3 liters or surgeon dissatisfaction), NMBA are used. This define the secondary use of NMBA.

Methods :

Anesthesia will be induced in all patients by target controlled infusions of propofol and sufentanil respectively with initial targets of 6 microgram/ml and 0,4 ng/ml.

The initial NMBA bolus in the NMBA group is 0,15 mg/kg of cisatracurium. A similar volume of isotonic saline serum is used in the placebo group.

The abdomen is inflated to 5, 10 and 15 mmHg and volumes at each pressure level are measured in order to evaluate the abdominal compliance.

After those measures, the anesthesiologist is unblinded of NMBA use. If the workspace volume is lesser than 3 liters, or, in case of surgeon dissatisfaction (using the surgical rating scale), NMBA can be used, defining secondary NMBA used.

Anesthesia is maintained by continous infusions of propofol and sufentanil aiming BIS target of 40 to 60.

When used, curarisation is maintained by a continuous infusion of cisatracurium (0,06 to 0,12 mg/kg/h) targetting 0 or 1 TOF response.

Safety issues : During anesthesia induction, if ventilation or tracheal intubation difficulties were to happen, the anesthesiologist is unblinded and any anesthesia protocol can be used.

ELIGIBILITY:
Inclusion Criteria:

* elective abdominal laparoscopy (cholecystectomy, colectomy, gastric bypass, sleeve gastrectomy, hepatic resection, splenectomy, hernial surgery, explorative laparoscopy)
* >18 yo
* patients who accept the protocol and sign it
* patients affiliated at the social security

Exclusion Criteria:

* formal indication of NMBA use (predictive difficult tracheal intubation, predictive difficult facial ventilation)
* patients who needs a crush induction
* NMBA allergia
* patients who present a contraindication to the propofol or sufentanil
* pregnancy
* breastfeeding womens
* patients protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Volume of pneumoperiteum laparoscopic workspace | Day 0 (after anesthesia induction)
  laparoscopic workspace assessed by volume of pneumoperiteum > 3 Liters
score SRS (Surgical Rating Scale) | Day 0 (after anesthesia induction)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France